CLINICAL TRIAL: NCT03267836
Title: A Phase Ib Study of Neoadjuvant Avelumab and Hypofractionated Proton Radiation Therapy Followed by Surgery for Recurrent Radiation-refractory Meningioma
Brief Title: Neoadjuvant Avelumab and Hypofractionated Proton Radiation Therapy Followed by Surgery for Recurrent Radiation-refractory Meningioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study sponsor wanted to terminate enrollment.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201711195
Record Dates: First submitted 2017-08-29; First posted 2017-08-30 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Meningioma; Meningioma, Adult
MeSH Terms: conditions — Meningioma | interventions — avelumab; Proton Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Avelumab + Proton Therapy (Experimental): * Avelumab will be started concurrently with proton therapy (up to 3 days before or after is permissible) and administered every 2 weeks for 3 months
  * Proton therapy 20 CGE (cobalt gray equivalent) will be given over 5 daily fractions of 4 CGE per day during weekdays
  * After 3 months of avelumab, patient will have a brain MRI evaluation, and radiological response will be assigned based on the iRANO criteria. Surgery will be performed as per routine clinical care
  * If the brain MRI after 3 months of avelumab shows complete response with no signs of residual tumor, no surgery will be indicated, and the patient may continue to take adjuvant avelumab for an additional 3 months.
  * After the patient has recovered from the surgery and if deemed medically eligible by the treating physician to receive additional immunotherapy, avelumab will be restarted and administered every 2 weeks for an additional 3 months
  Interventions: Drug: Avelumab; Radiation: Proton Therapy; Procedure: Surgery

INTERVENTIONS:
Drug: Avelumab — -10mg/kg IV
  Other Names: Bavencio
Radiation: Proton Therapy — -Proton therapy will start concurrently with the first dose of avelumab (up to 3 days before or after is permissible) and will be administered once daily during weekdays (Monday through Friday).
Procedure: Surgery — -Standard of care

SUMMARY:
Meningioma is the most common central nervous system (CNS) tumor and accounts for approximately 30% of all CNS tumors. For meningioma recurring after surgery and radiation therapy, there is no effective medical therapy. Repeat surgery or radiation therapy may be possible, but they are temporizing measures with limited durable relief. PD-L1 expression in meningioma is increased for recurrent tumors or prior radiation therapy, and a recent case study reported significant reduction of an intracranial meningioma after 6 months of PD-L1 blockade. Radiation has been shown to augment immune response when combined with PD-L1 blockade. Proton radiation therapy has higher relative biological effectiveness (RBE) and may further amplify the above immunological signals. Combination of proton radiation therapy administered concurrently with PD-L1 inhibitor may maximize immune response for recurrent meningioma. However, confirmation of the increased immunogenicity or increased tumor infiltrating lymphocytes using the combination of radiation therapy and PD-L1 blockade have not been confirmed in patients. The proposed study will be a single institution, single-arm, open-label, phase Ib study to combine neoadjuvant avelumab (a PD-L1 inhibitor) with hypofractionated proton therapy of 20 CGE (cobalt gray equivalent) over 5 fractions followed by planned surgery for recurrent radiation-refractory meningioma. This study is designed to provide proof of concept to demonstrate on-target effect of the combination to increase immunogenicity by directly examining the resected tumor for immune response and to evaluate preliminary clinical efficacy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent or progressive histologically confirmed WHO grade I-III meningioma which has failed maximal safe resection and radiation therapy.
* At least one prior surgery with available archival formalin-fixed paraffin-embedded (FFPE) tumor blocks. In the case that tumor block is unavailable, unstained tissue sections may be used in its place.
* Prior treatment must include external beam radiation, radiosurgery, or combination of both.
* Deemed eligible for additional partial resection by treating physician and determined to be safe to receive 3 months of neoadjuvant therapy before planned surgery.
* Age ≥ 18 years old. 6. Karnofsky performance status (KPS) ≥ 60.
* Adequate organ and bone marrow function (as defined by the following laboratory values):

  * Absolute neutrophil count ≥ 1.5 × 10⁹ cells per L
  * Platelet count ≥ 100 × 10⁹ platelets per L
  * Hemoglobin ≥ 9 g/dL but transfusion allowed
  * Total bilirubin concentration of ≤ 1.5 × the upper limit of normal [ULN] range
  * Aspartate aminotransferase and alanine aminotransferase concentrations of ≤ 2.5 × ULN)
  * Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula.
* Dexamethasone dose ≤ 4mg daily.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in the study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB approved written informed consent document (or legally authorized representative, if applicable)

Exclusion Criteria:

* Previous treatment with PD-1 or PD-L1 directed therapy.
* Active infection requiring systemic therapy.
* Uncontrolled intercurrent illness including, but not limited to, clinically significant (i.e. active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), congestive heart failure (≥ NYHA class II), unstable angina pectoris, or serious cardiac arrhythmia requiring medication.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive).
* Currently receiving any other investigational agents.
* Current use of immunosuppressive medication, EXCEPT for the following:

  * Intranasal, inhaled, topical steroids, or local steroid injection (e.g. intra-articular injection)
  * Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication)
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
* Prior organ transplantation including allogeneic stem cell transplantation.
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis, or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines.
* History of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition to avelumab or other agents used in the study (or monoclonal antibodies).
* Persisting toxicity related to prior therapy (CTCAE > grade 1); however, alopecia, sensory neuropathy ≤ grade 2, or other ≤ grade 2 not constituting a safety risk based on the investigator's judgment are acceptable.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Immunogenicity as measured by changes of CD8+/CD4+ tumor infiltrating lymphocytes (TILs) in recurrent radiation-refractory meningioma | Through time of progression (up to 6 months after completion of treatment - estimated to be 12 months)
  -The change of CD8+/CD4+ TILs in the tumor specimens over time will be compared using paired t-test or Wilcoxon rank-sum test as appropriate and plotted using the box plot. The association between TILs increase and clinical response will also be explored by comparing the differences in theses biomarkers between responders versus non-responders using t-test or Mann-Whitney rank-sum test as appropriate.

SECONDARY OUTCOMES:
Safety of proton therapy and avelumab in combination as measured by The number and percentage of subjects experiencing each type of adverse event will be tabulated by severity, and relationship to treatment. | 6 months after completion of treatment (estimated to be 12 months)
  If appropriate, confidence intervals will be used to characterize the precision of the estimate.
Radiological response | 3 months of immunotherapy
  * 95% confidence intervals will be calculated
  * Response and progression will be evaluated in this study using the modified updated response assessment criteria for high-grade gliomas: Response Assessment in Neuro-Oncology (RANO) working group guideline
Pathologic response | 3 months of immunotherapy
  -Will be evaluated by board-certified neuropathologist on formalin-fixed paraffin-embedded tumor specimens stained with hematoxylin and eosin, where responders are defined as ≥30% necrosis/reactive changes and ≤50% viable tumor.
Progression-free survival (PFS) | Through 2 years after completion of treatment (estimated to be 2.5 years)
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Median PFS and their 95% confidence intervals will be assessed using Kaplan-Meier product limit methods.
Overall survival (OS) | Through 2 years after completion of treatment (estimated to be 2.5 years)
  -Median OS and their 95% confidence intervals will be assessed using Kaplan-Meier product limit methods.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Huang, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu